CLINICAL TRIAL: NCT05725655
Title: Hot Water Immersion in Rehabilitation After Myocardial Infarction (HOT-MI) - a Randomized Controlled Study
Brief Title: Hot Water Immersion After Myocardial Infarction
Acronym: HOT-MI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 279938
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Cardiac Disease; Cardiac Rehabilitation
MeSH Terms: conditions — Heart Diseases | interventions — Hyperthermia, Induced

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hot water immersion (Experimental): Patients allocated to hot water immersion will enter a bath and submerge down to the neck in warm water (40 degrees celsius) for 20 min.
  Interventions: Other: Thermotherapy
- Control (No Intervention): Patients allocated to control group will sit down for a 20 min rest.

INTERVENTIONS:
Other: Thermotherapy — Hot baths directly after an exercise session
  Arms: Hot water immersion

SUMMARY:
Myocardial infarction (MI) is a leading cause of death in developed countries, including Sweden. Standard treatment for patients after MI includes exercise-based cardiac rehabilitation which contributes to improved cardiovascular function and reduces the risk of hospital readmissions, new cardiovascular events and mortality. Thermotherapy may also have beneficial effects on cardiovascular disease by a reduction in inflammatory status and improved metabolism and vascular function. Given the well-documented effects of exercise training on cardiac rehabilitation and recent evidence that thermotherapy may improve cardiovascular function, we wish to investigate the effect of exercise combined with hot water immersion (HWI) in cardiac rehabilitation post-MI.

This is a single-centre, randomized controlled clinical trial in patients with recent MI. Our aim is to investigate whether exercise training combined with HWI improves inflammatory and metabolic status, cardiovascular function as well as psychological well-being, compared with exercise training alone. Patients will be randomized 1:1 to an 8 week intervention with exercise training 2 times per week followed by 15 minutes of hot water immersion, or to a control group with exercise training alone. The primary endpoint is changes in the inflammatory marker interleukin (IL-) 6 between groups at 8 weeks. Secondary endpoints include other biomarkers of inflammation, metabolism, effects on cardiovascular function and psychological benefits.

Secondary prevention after MI has improved during the last decades but readmissions and death following acute MI remain large health challenges. If HWI in addition to standard cardiac rehabilitation can lower inflammation more than standard therapy alone, and improve metabolic, cardiovascular and psychological status, it could be a cost-effective and safe complementary strategy for secondary prevention after MI, particularly for those with limited exercise capability.

ELIGIBILITY:
Inclusion criteria

* Patients with a diagnosis of ST-elevation myocardial infarction (STEMI) or non-STEMI
* Concomitant participation in standard care exercise-based cardiac rehabilitation
* Male or female patients ≥ 18 years
* Written informed consent

Exclusion criteria

* Regularly performing hot water immersion, sauna or other types of thermotherapy
* Not willing to perform hot water immersion regularly
* Febrile illness or acute, ongoing infection
* <18 years of age
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Concentrations of interleukin 6 (IL-6) in blood | 8 weeks (aiming at 16 bath (or control) sessions during the intervention period
  Change in IL-6 between groups after 8 weeks of intervention (aiming at 16 bath (or control) sessions during the intervention period)

SECONDARY OUTCOMES:
Concentrations of other biomarkers of inflammation in blood | 8 weeks
  Change in IL -1b, IL-10, tumor necrosis factor (TNF)-a, High sensitivity C-reactive protein, heat shock protein-72 after 8 weeks of intervention
Concentrations of biomarkers of metabolism in blood | 8 weeks
  Heat shock factor (HSF)-1, High density lipoprotein, Low density lipoprotein, triglycerides, cholesterol, leptin and adiponectin, glucose, insulin
Change in percent in endothelial flow-mediated dilatation (FMD) | 8 weeks
  Change after 8 weeks of intervention
Change in sympathetic/parasympathetic activity | 8 weeks
  Change in heart rate variability after 8 weeks of intervention
Change in score of participants´ subjectively reported psychological well-being | 8 weeks
  Measured with the Questionnaire Clinical Outcomes in Routine Evaluation (Core-GP), change after 8 weeks of intervention
Change in diastolic and systolic blood pressure (mm(Hg) | 8 weeks
  Change after 8 weeks of intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Örebro University hospital, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No